CLINICAL TRIAL: NCT02687841
Title: A Uremic Toxin Absorbent (AST-120) to Treat Hospital Acquired Acute Kidney Injury - A Open Label Randomized Control Trial
Brief Title: A Uremic Toxin Absorbent (AST-120) to Treat Hospital Acquired Acute Kidney Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); National Taiwan University Hospital Hsin-Chu Branch (Other); China Medical University Hospital (Other); Taoyuan General Hospital (Other Government); Taipei Medical University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, KWAN-DUN WU MD. PhD., National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201502003MIPB
Record Dates: First submitted 2016-01-26; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; indoxylsulfate; p-cresol; AST-120
MeSH Terms: conditions — Acute Kidney Injury | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AST-120 and PTX (Experimental): AST-120 2g 4 times a day for 5 days then AST-120 2g 3 times a day for 5 days Pentapentoxifylline 400mg QD for 10 days
  Interventions: Drug: AST-120and pentoxyphylline (PTX)
- PTX (Active Comparator): Pentapentoxifylline 400mg QD for 10 days
  Interventions: Drug: pentoxyphylline (PTX)

INTERVENTIONS:
Drug: AST-120and pentoxyphylline (PTX) — AST-120 2g 4 times a day for 5 days then AST-120 2g 3 times a day for 5 days pentoxyphylline 400mg QD PO x 10 days.
  Arms: AST-120 and PTX
Drug: pentoxyphylline (PTX) — pentoxyphylline 400mg QD PO x 10 days.
  Arms: PTX

SUMMARY:
Hospital acquired acute kidney injury is an important negative outcome predictor for hospitalized patients. Uremic toxins accumulated after a given renal insult. Some of these uremic toxins are protein bound and may accumulated after renal impairment, owing to both impaired filtration, and inflammation. Recent animal studies have reported that accumulation of uremic toxins, namely indoxyl sulfate and p-cresol, would down regulate endothelial progenitor cells and in turn affect renal recovery. Elimination of these protein bound uremic toxins with an activated charcoal would help restore endothelial function. We will conduct a double blinded randomized placebo controlled trial, which aims to determine that if oral activated charcoal will retard progression of AKI. Also, a panel of markers for endothelial function will also be determined.

ELIGIBILITY:
This is a prospective randomized placebo controlled trial. All patients admitted to participating centers with newly diagnosed acute kidney injury (AKI) will be screened for eligibility. The diagnosis of AKI will be determined and staged according to the KIGO-AKI Guideline.11 The inclusion criteria include:

1. Age ≥ 20 years old on the day of admission
2. AKI develops during admission, as defined with KDIGO-AKI Guideline,11 namely, elevation of serum creatinine above 0.3mg/dL within two days, above 1.5times baseline.

Patients with the following conditions will be excluded:

1. Baseline estimated glomerular filtration rates (eGFR) less than 30ml/min/1.73m2 or greater than 90ml/min/1.73m2 according to MDRD equation.
2. Acute kidney injury diagnosed in the indexed admission (according to baseline creatinine)
3. Ileus or under fasting status
4. Previous gastrointestinal operation.
5. Chronic constipation, as defined with bowel movement less than three times a day. If usage of oral laxatives can achieve bowel movement of more than 3 times a day, this patient will not be excluded.
6. Patients had ever undergone any modality of renal replacement therapy (RRT)
7. Patients with major hemorrhage, as defined with requirement of blood transfusion during index admission.
8. Patients with a biopsy proved or clinically diagnosed liver cirrhosis, Child classification B or C.
9. Patients with a congestive heart failure of NYHA Class III or IV, or requirement of inotropic agents.
10. Patients with a chronic lung disease requiring non-invasive or invasive positive pressure ventilation.
11. Solid organ or hematological transplantation donors.
12. Patients who had been diagnosed as AKI in the index hospitalization, as defined with KDIGO 2012 criteria.
13. Patients with oliguric acute kidney injury, as defined with less than 500cc/day.
14. Evidence of obstructive acute kidney injury under kidney echosonography.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Total recovery of kidney function, which is defined as less than 1.5 times pre-morbid creatinine levels on the 10th day of intervention. | 10 days

SECONDARY OUTCOMES:
Total recovery of serum creatinine on Day 5 | 5 days
  defined with less than 1.5 times elevation of pre-morbid plasma creatinine level.
Needing renal replacement therapy on day 10. | 10 days
Degree of serum creatinine elevation | 10 days
  as calculated with ratios between highest serum creatinine and pre-morbid creatinine during study period
The degree of Indoxyl sulfate change on Day 10 (%) | 10 days
The degree of Indoxyl sulfate change on Day 5 (%) | 5 days
The degree of p-cresol change on Day 10 (%) | 10 days
The degree of p-cresol change on Day 5 (%) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: YU-SHENG WU, Principal Investigator — National Taiwan University Hospital; Tao-Min Huang, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch; Wei-Shun Yang, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch; JUI-HSIANG LIN, Principal Investigator — Taoyuan General Hospital; Ya-Fei Yang, Principal Investigator — China Medical University Hospital; Chan-Yu Lin, Principal Investigator — Chang Gung Memorial Hospital; Heng-Chih Pan, Principal Investigator — Chang Gung Memorial Hospital; Chih-Chin Kao, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- National Taiwan University Hospital Yun-Lin Branch, Douliu, Taiwan, Taiwan